CLINICAL TRIAL: NCT00170950
Title: A Prospective, Multinational, Multicenter Trial to Compare the Effects of Amlodipine/Benazepril to Benazepril and Hydrochlorothiazide Combined on the Reduction of Cardiovascular Morbidity and Mortality in Patients With High Risk Hypertension
Brief Title: Avoiding Cardiovascular Events Through Combination Therapy in Patients Living With Systolic Hypertension
Acronym: ACCOMPLISH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early because of significant efficacy results for the primary endpoint in favor of benazepril/amlodipine treatment.
Sponsor: Novartis (Industry)
Responsible Party: Study Diorector, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCIB002I2301; NCT00097864 (obsolete NCT alias)
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Hypertension
Keywords: cardiovascular morbidity; cardiovascular mortality; benazepril; amlodipine; high risk population
MeSH Terms: conditions — Hypertension | interventions — benazepril; Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Benazepril/amlodipine (Experimental): Patients were instructed to take one capsule with water in the morning, except on the morning of their next office visit. On office visit days, study medication was taken after completion of the visit evaluations. Following randomization, all patients were treated at Dose Level 1 for 4 weeks, followed by a forced titration to Dose Level 2 for a subsequent 4 week period. Thereafter, patients were titrated as needed to Dose Level 3 to achieve a target blood pressure of < 140/< 90 mm Hg. For patients with diabetes or chronic kidney disease, investigators were encouraged to use a target blood pressure of 130/80 mm Hg.
  Interventions: Drug: Benazepril/amlodipine 20/5 mg - Dose Level 1 from Day 1 to Month 1; Drug: Benazepril/amlodipine 40/5 mg - Dose Level 2 from Month 1 to Month 2; Drug: Benazepril/amlodipine 40/10 mg - Dose Level 3 from Month 2 to Month 3 and thereafter
- Benazepril/hydrochlorothiazide (Active Comparator): Patients were instructed to take one capsule with water in the morning, except on the morning of their next office visit. On office visit days, study medication was taken after completion of the visit evaluations. Following randomization, all patients were treated at Dose Level 1 for 4 weeks, followed by a forced titration to Dose Level 2 for a subsequent 4 week period. Thereafter, patients were titrated as needed to Dose Level 3 to achieve a target blood pressure of < 140/< 90 mm Hg. For patients with diabetes or chronic kidney disease, investigators were encouraged to use a target blood pressure of 130/80 mm Hg.
  Interventions: Drug: Benazepril/hydrochlorothiazide 20/12.5 mg - Dose Level 1 from Day 1 to Month 1; Drug: Benazepril/hydrochlorothiazide 40/12.5 mg - Dose Level 2 from Month 1 to Month 2; Drug: Benazepril/hydrochlorothiazide 40/25 mg - Dose Level 3 from Month 2 to Month 3 and thereafter

INTERVENTIONS:
Drug: Benazepril/amlodipine 20/5 mg - Dose Level 1 from Day 1 to Month 1 — Benazepril hydrochloride (HCl)/amlodipine besylate 10/5 mg capsules for oral administration once daily.
  Arms: Benazepril/amlodipine
Drug: Benazepril/amlodipine 40/5 mg - Dose Level 2 from Month 1 to Month 2 — Benazepril hydrochloride (HCl)/amlodipine besylate 20/5 mg capsules for oral administration once daily.
  Arms: Benazepril/amlodipine
Drug: Benazepril/amlodipine 40/10 mg - Dose Level 3 from Month 2 to Month 3 and thereafter — Benazepril hydrochloride (HCl)/amlodipine besylate: 40/10 mg capsules for oral administration once daily. Patients titrated to this dose level had the possibility of subsequent free add-on antihypertensive agents after month 3 based on target blood pressure.
  Arms: Benazepril/amlodipine
Drug: Benazepril/hydrochlorothiazide 20/12.5 mg - Dose Level 1 from Day 1 to Month 1 — Benazepril hydrochloride (HCl)/hydrochlorothiazide (HCTZ) 20/12.5 mg capsules for oral administration once daily.
  Arms: Benazepril/hydrochlorothiazide
Drug: Benazepril/hydrochlorothiazide 40/12.5 mg - Dose Level 2 from Month 1 to Month 2 — Benazepril hydrochloride (HCl)/hydrochlorothiazide (HCTZ) 40/12.5 mg capsules for oral administration once daily.
  Arms: Benazepril/hydrochlorothiazide
Drug: Benazepril/hydrochlorothiazide 40/25 mg - Dose Level 3 from Month 2 to Month 3 and thereafter — Benazepril hydrochloride (HCl)/hydrochlorothiazide (HCTZ) 40/25 mg capsules for oral administration once daily. Patients titrated to this dose level had the possibility of subsequent free add-on antihypertensive agents after month 3 based on target blood pressure.
  Arms: Benazepril/hydrochlorothiazide

SUMMARY:
A comparison study of two combination drugs, amlodipine/benazepril and benazepril/HCTZ to evaluate the effectiveness of the combination on reducing heart disease and death in a high risk hypertensive population.

ELIGIBILITY:
Inclusion Criteria:

* At least 55 years of age.
* Previously untreated or treated hypertension.
* For patients >= 60 years, evidence of at least one CV disease or target organ damage, or for patients 55-59 years evidence of at least two CV diseases or target organ damage from two different organ systems as defined in the protocol.

Exclusion Criteria:

* Allergy to any of the drugs administered in this trial.
* Current angina pectoris (ie, no anginal event requiring NTG within 1 month prior to Visit 1).
* Secondary hypertension.
* Refractory hypertension defined as SBP >= 180 mmHg and/or DBP >= 110 mmHg unresponsive to triple-drug regimens of sympatholytics, diuretics and vasodilators.
* History of symptomatic heart failure (NYHA classes II-IV) or ejection fraction < 40%.
* Myocardial infarction, coronary revascularization (CABG or PCI), unstable angina within one month of Visit 1.
* Stroke or transient ischemic event (TIA) within 3 months of Visit 1.
* Significant obstructive valvular cardiovascular disease or any valvular disease expected to lead to surgery during the course of the study.
* Evidence of hepatic disease (AST or ALT values >= 2 X upper limit of normal).
* Impaired renal function (serum creatinine >= 2.5 mg/dL (221 µmol/L)).
* Baseline serum potassium of > 5.2 meq/L not on potassium supplements.
* History of malignancy including leukemia and lymphoma (but not basal cell skin cancer) within the last 5 years.
* History of clinically significant auto immune disorders such as Systemic Lupus Erythematosus.
* Significant non-cardiovascular illness or condition likely to result in death prior to trial completion, e.g., major organ transplant (life expectancy <5 years).
* Significant cardiovascular disease such as an aortic aneurysm ≥ 6 cm, likely requiring surgical intervention during the course of the study.

Other protocol-defined exclusion criteria applied to the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11506 (Actual)
Dates: Start 2003-10; Primary Completion 2008-01 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (5):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- sites in Denmark, Denmark, Denmark
- sites in Finland, Finland, Finland
- sites in Norway, Norway, Norway
- sites in Sweden, Sweden, Sweden

REFERENCES:
- [Result] Jamerson K, Weber MA, Bakris GL, Dahlof B, Pitt B, Shi V, Hester A, Gupte J, Gatlin M, Velazquez EJ; ACCOMPLISH Trial Investigators. Benazepril plus amlodipine or hydrochlorothiazide for hypertension in high-risk patients. N Engl J Med. 2008 Dec 4;359(23):2417-28. doi: 10.1056/NEJMoa0806182. PMID 19052124
- [Derived] Brook RD, Kaciroti N, Bakris G, Dahlof B, Pitt B, Velazquez E, Weber MA, Jamerson KA. Cardiovascular Benefits of Angiotensin-Converting Enzyme Inhibition Plus Calcium Channel Blockade in Patients Achieving Tight Blood Pressure Control and With Resistant Hypertension. Am J Hypertens. 2021 May 22;34(5):531-539. doi: 10.1093/ajh/hpaa192. PMID 33216879
- [Derived] Weber MA, Jamerson K, Bakris GL, Weir MR, Zappe D, Zhang Y, Dahlof B, Velazquez EJ, Pitt B. Effects of body size and hypertension treatments on cardiovascular event rates: subanalysis of the ACCOMPLISH randomised controlled trial. Lancet. 2013 Feb 16;381(9866):537-45. doi: 10.1016/S0140-6736(12)61343-9. Epub 2012 Dec 6. PMID 23219284
- [Derived] Weber MA, Bakris GL, Jamerson K, Weir M, Kjeldsen SE, Devereux RB, Velazquez EJ, Dahlof B, Kelly RY, Hua TA, Hester A, Pitt B; ACCOMPLISH Investigators. Cardiovascular events during differing hypertension therapies in patients with diabetes. J Am Coll Cardiol. 2010 Jun 29;56(1):77-85. doi: 10.1016/j.jacc.2010.02.046. PMID 20620720
- [Derived] Bakris GL, Sarafidis PA, Weir MR, Dahlof B, Pitt B, Jamerson K, Velazquez EJ, Staikos-Byrne L, Kelly RY, Shi V, Chiang YT, Weber MA; ACCOMPLISH Trial investigators. Renal outcomes with different fixed-dose combination therapies in patients with hypertension at high risk for cardiovascular events (ACCOMPLISH): a prespecified secondary analysis of a randomised controlled trial. Lancet. 2010 Apr 3;375(9721):1173-81. doi: 10.1016/S0140-6736(09)62100-0. Epub 2010 Feb 18. PMID 20170948

RESULTS

PARTICIPANT FLOW:
Groups:
- Benazepril/Amlodipine: Benazepril hydrochloride (HCl)/amlodipine besylate: 20/5 mg (Dose Level 1 from Day 1 to Month 1), 40/5 mg (Dose Level 2 from Month 1 to Month 2), and 40/10 mg (Dose Level 3 from Month 2 to Month 3 and thereafter) capsules for oral administration once daily
- Benazepril/Hydrochlorothiazide: Benazepril hydrochloride (HCl)/hydrochlorothiazide (HCTZ): 20/12.5 mg (Dose Level 1 from Day 1 to Month 1), 40/12.5 mg (Dose Level 2 from Month 1 to Month 2), and 40/25 mg (Dose Level 3 from Month 2 to Month 3 and thereafter) capsules for oral administration once daily
Period: Overall Study
Arm/Group | Benazepril/Amlodipine | Benazepril/Hydrochlorothiazide
Started | 5744 | 5762
Completed | 4859 | 4852
Not Completed | 885 | 910
Not completed — Death | 236 | 274
Not completed — Withdrawal by Subject | 496 | 498
Not completed — Lost to Follow-up | 134 | 115
Not completed — Missing | 2 | 1
Not completed — Termination Data Not Recorded | 17 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benazepril/Amlodipine | Benazepril/Hydrochlorothiazide | Total
Number analyzed (Participants) | 5744 | 5761 | 11505
Age, Continuous [Mean (Standard Deviation); unit: Years] — Demographic data for 1 patient in the benazepril/hydrochlorothiazide was not available.
  Years | 68.4 (6.86) | 68.3 (6.86) | 68.4 (6.86)
Sex: Female, Male [Count of Participants; unit: Participants] — Demographic data for 1 patient in the benazepril/hydrochlorothiazide was not available.
  Participants
    Female | 2296 | 2246 | 4542
    Male | 3448 | 3515 | 6963

OUTCOME MEASURES:

1. Primary Outcome: Time-to-event Analysis of Percentage of Patients With a Composite Cardiovascular (CV) Morbidity or Mortality Event
Description: CV morbidity was defined as non-fatal myocardial infarction (MI), non-fatal stroke, hospitalization for unstable angina, resuscitated sudden death, or coronary revascularization procedure. CV mortality was defined as death due to MI, stroke, coronary intervention, congestive heart failure (CHF), sudden cardiac death, or other CV causes.
Time Frame: For each patient, baseline to time of first CV morbidity or mortality event (or last exposure if no event occurred). (Median duration of exposure was 33.4 months. [25th to 75th percentiles: 21 to 41 months.])
Population: Intent-to-treat population: All randomized patients by assigned treatment group
Measure: Number; unit: Percentage of Patients with an event
Arm/Group | Benazepril/Amlodipine | Benazepril/Hydrochlorothiazide
Number analyzed (Participants) | 5744 | 5762
Percentage of Patients with an event | 9.6 | 11.8

2. Secondary Outcome: Time-to-event Analysis of Percentage of Patients With a Composite Cardiovascular (CV) Morbidity Event
Description: Cardiovascular morbidity was defined as including any of the following events: non-fatal MI, non-fatal stroke, hospitalization for unstable angina, resuscitated sudden death, or coronary revascularization procedure (PCI or CABG).
Time Frame: For each patient, baseline to time of first CV morbidity event (or last exposure if no event occurred). (Median duration of exposure was 33.4 months. [25th to 75th percentiles: 21 to 41 months.])]
Population: Intent-to-treat population: All randomized patients by assigned treatment group
Measure: Number; unit: Percentage of Patients with an Event
Arm/Group | Benazepril/Amlodipine | Benazepril/Hydrochlorothiazide
Number analyzed (Participants) | 5744 | 5762
Percentage of Patients with an Event | 8.6 | 10.3

3. Secondary Outcome: Time-to-event Analysis of Percentage of Patients With a Cardiovascular (CV) Mortality Event, Non-fatal Myocardial Infarction (MI), or Non-fatal Stroke
Description: CV mortality was defined as death due to sudden cardiac death, fatal MI, fatal stroke, coronary intervention, congestive heart failure (CHF), or other CV causes.
Time Frame: For each patient, baseline to time of first CV mortality event, MI (non-fatal), or stroke (non-fatal) (or last exposure if no event occurred). (Median duration of exposure was 33.4 months. [25th to 75th percentiles: 21 to 41 months.])
Population: Intent-to-treat population: All randomized patients by assigned treatment group
Measure: Number; unit: Percentage of Patients with an Event
Arm/Group | Benazepril/Amlodipine | Benazepril/Hydrochlorothiazide
Number analyzed (Participants) | 5744 | 5762
Percentage of Patients with an Event | 5.0 | 6.3

ADVERSE EVENTS:
Time Frame: Double-blind period
Description: Safety population includes all randomized patients who took at least one dose of study medication by actual treatment group (7 Benazepril / Amlodipine and 2 Benazepril / HCTZ patients did not take study medication; 3 patients assigned to Benazepril / HCTZ received Benazepril / Amlodipine medication instead).
Groups:
- Benazepril / Amlodipine: Benazepril hydrochloride (HCl)/amlodipine besylate: 20/5 mg (Dose Level 1), 40/5 mg (Dose Level 2), and 40/10 mg (Dose Level 3) capsules for oral administration once daily
- Benazepril / HCTZ: Benazepril hydrochloride (HCl)/hydrochlorothiazide (HCTZ): 20/12.5 mg (Dose Level 1), 40/12.5 mg (Dose Level 2), and 40/25 mg (Dose Level 3) capsules for oral administration once daily
Arm/Group | Benazepril / Amlodipine | Benazepril / HCTZ
Serious Adverse Events (participants affected / at risk) | 1844/5740 | 2026/5757
Other Adverse Events (participants affected / at risk) | 3077/5740 | 2663/5757
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Benazepril / Amlodipine (N=5740) | Benazepril / HCTZ (N=5757)
Acquired haemophilia (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 34 | 41
Blood disorder (Blood and lymphatic system disorders) | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 2
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 | 2
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 | 1
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 | 3
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Thrombocythaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
AV dissociation (Cardiac disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 5 | 9
Acute myocardial infarction (Cardiac disorders) | 17 | 11
Angina pectoris (Cardiac disorders) | 85 | 106
Angina unstable (Cardiac disorders) | 113 | 131
Aortic valve disease (Cardiac disorders) | 1 | 2
Aortic valve incompetence (Cardiac disorders) | 1 | 3
Aortic valve stenosis (Cardiac disorders) | 3 | 1
Arrhythmia (Cardiac disorders) | 6 | 8
Arteriosclerosis coronary artery (Cardiac disorders) | 14 | 12
Atrial fibrillation (Cardiac disorders) | 115 | 113
Atrial flutter (Cardiac disorders) | 7 | 8
Atrial tachycardia (Cardiac disorders) | 0 | 2
Atrioventricular block (Cardiac disorders) | 3 | 1
Atrioventricular block complete (Cardiac disorders) | 5 | 4
Atrioventricular block first degree (Cardiac disorders) | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 4 | 3
Bradyarrhythmia (Cardiac disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 21 | 31
Bundle branch block left (Cardiac disorders) | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 6 | 14
Cardiac discomfort (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 8 | 16
Cardiac failure congestive (Cardiac disorders) | 99 | 86
Cardiac hypertrophy (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardiac ventricular disorder (Cardiac disorders) | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 5 | 3
Cardiogenic shock (Cardiac disorders) | 3 | 3
Cardiomegaly (Cardiac disorders) | 1 | 2
Cardiomyopathy (Cardiac disorders) | 3 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 2
Congestive cardiomyopathy (Cardiac disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 112 | 124
Coronary artery insufficiency (Cardiac disorders) | 1 | 2
Coronary artery occlusion (Cardiac disorders) | 7 | 18
Coronary artery restenosis (Cardiac disorders) | 0 | 2
Coronary artery stenosis (Cardiac disorders) | 16 | 21
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 4
Left ventricular dysfunction (Cardiac disorders) | 0 | 2
Mitral valve incompetence (Cardiac disorders) | 3 | 2
Myocardial infarction (Cardiac disorders) | 91 | 126
Myocardial ischaemia (Cardiac disorders) | 10 | 13
Palpitations (Cardiac disorders) | 3 | 3
Pericardial effusion (Cardiac disorders) | 3 | 2
Pericarditis (Cardiac disorders) | 2 | 1
Right ventricular failure (Cardiac disorders) | 3 | 1
Sick sinus syndrome (Cardiac disorders) | 15 | 20
Sinus arrest (Cardiac disorders) | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 2 | 1
Sinus bradycardia (Cardiac disorders) | 3 | 3
Sinus tachycardia (Cardiac disorders) | 2 | 1
Supraventricular tachycardia (Cardiac disorders) | 3 | 5
Tachyarrhythmia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 4 | 8
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1
Trifascicular block (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 3 | 1
Ventricular hypokinesia (Cardiac disorders) | 1 | 0
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 10 | 10
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Congenital syphilitic osteochondritis (Congenital, familial and genetic disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 2
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 11 | 9
Vertigo positional (Ear and labyrinth disorders) | 2 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Adrenal mass (Endocrine disorders) | 1 | 1
Antidiuretic hormone abnormality (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 2 | 2
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 3 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 2
Thyroid mass (Endocrine disorders) | 2 | 1
Entropion (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 1
Eyelid ptosis (Eye disorders) | 1 | 0
Hyphaema (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 2 | 0
Retinal detachment (Eye disorders) | 0 | 1
Retinal tear (Eye disorders) | 1 | 0
Retinal vein thrombosis (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 2 | 2
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 21 | 20
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 9 | 12
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 2
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1
Caecitis (Gastrointestinal disorders) | 2 | 1
Colitis (Gastrointestinal disorders) | 7 | 8
Colitis ischaemic (Gastrointestinal disorders) | 6 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1
Colonic fistula (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 2 | 2
Colonic stenosis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 2
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1
Diabetic gastropathy (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 17 | 20
Diverticulum (Gastrointestinal disorders) | 4 | 5
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 | 2
Diverticulum oesophageal (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 4 | 5
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 3
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 5
Enterocele (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 3 | 2
Faecal incontinence (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 1
Food poisoning (Gastrointestinal disorders) | 2 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 4 | 6
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 3
Gastritis (Gastrointestinal disorders) | 14 | 17
Gastritis erosive (Gastrointestinal disorders) | 2 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 35 | 29
Gastrointestinal necrosis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 14
Gastrooesophagitis (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 2 | 5
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 3 | 2
Ileus (Gastrointestinal disorders) | 2 | 8
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 2 | 3
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 7 | 8
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal infarction (Gastrointestinal disorders) | 2 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 2
Intestinal mass (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 5 | 4
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 2 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 3 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 | 5
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 5
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 9 | 18
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Oesophageal disorder (Gastrointestinal disorders) | 0 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal rupture (Gastrointestinal disorders) | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 3 | 1
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 16 | 23
Pancreatitis acute (Gastrointestinal disorders) | 6 | 8
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 3 | 3
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 5 | 5
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 2
Retching (Gastrointestinal disorders) | 1 | 0
Retroperitoneal fibrosis (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 7 | 7
Tongue oedema (Gastrointestinal disorders) | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 2 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 2 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 9
Volvulus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 13 | 13
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 9 | 16
Cardiac death (General disorders) | 4 | 2
Catheter related complication (General disorders) | 0 | 2
Catheter site haematoma (General disorders) | 0 | 1
Chest discomfort (General disorders) | 9 | 7
Chest pain (General disorders) | 35 | 40
Chills (General disorders) | 2 | 0
Death (General disorders) | 4 | 7
Decapitation (General disorders) | 1 | 0
Drowning (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 8
Gait disturbance (General disorders) | 3 | 2
General physical health deterioration (General disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Hernia (General disorders) | 3 | 2
Hernia obstructive (General disorders) | 0 | 1
Impaired healing (General disorders) | 3 | 2
Malaise (General disorders) | 1 | 1
Multi-organ failure (General disorders) | 3 | 1
Non-cardiac chest pain (General disorders) | 64 | 50
Oedema (General disorders) | 0 | 3
Oedema peripheral (General disorders) | 10 | 8
Pelvic mass (General disorders) | 1 | 2
Perforated ulcer (General disorders) | 1 | 0
Pyrexia (General disorders) | 7 | 7
Sudden cardiac death (General disorders) | 1 | 3
Sudden death (General disorders) | 6 | 10
Ulcer (General disorders) | 1 | 1
Vestibulitis (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 3
Biliary dilatation (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 12 | 21
Cholecystitis acute (Hepatobiliary disorders) | 7 | 9
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 5
Cholelithiasis (Hepatobiliary disorders) | 16 | 27
Cholestasis (Hepatobiliary disorders) | 0 | 1
Chronic hepatitis (Hepatobiliary disorders) | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 3
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 1
Hepatic congestion (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 2
Jaundice (Hepatobiliary disorders) | 1 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 0 | 1
Allergy to arthropod sting (Immune system disorders) | 1 | 2
Allergy to vaccine (Immune system disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 2
Food allergy (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 1
Sarcoidosis (Immune system disorders) | 1 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 3 | 0
Abscess intestinal (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 2 | 2
Abscess neck (Infections and infestations) | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 1
Amoebiasis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 6 | 9
Arthritis bacterial (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 1
Atypical mycobacterial infection (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 2
Bacterial sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 21 | 17
Bronchitis bacterial (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 2
Bursitis infective (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 39 | 22
Cellulitis orbital (Infections and infestations) | 0 | 1
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Cellulitis streptococcal (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 3 | 3
Clostridial infection (Infections and infestations) | 1 | 2
Clostridium difficile colitis (Infections and infestations) | 2 | 7
Coccidioidomycosis (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 1 | 0
Cystitis klebsiella (Infections and infestations) | 0 | 1
Dacryocystitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 5 | 2
Diabetic foot infection (Infections and infestations) | 0 | 1
Diabetic gangrene (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 6 | 14
Eczema infected (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Encephalitis herpes (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 2
Endocarditis bacterial (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 10 | 2
Escherichia infection (Infections and infestations) | 2 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 2 | 1
Febrile infection (Infections and infestations) | 0 | 3
Fungal skin infection (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 4 | 4
Gastroenteritis (Infections and infestations) | 15 | 30
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 1
Gastroenteritis shigella (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 10 | 7
Gastrointestinal infection (Infections and infestations) | 0 | 1
Graft infection (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 0 | 1
Groin infection (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 1
Helicobacter infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 4 | 1
Histoplasmosis (Infections and infestations) | 0 | 1
Infected epidermal cyst (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 3
Infection (Infections and infestations) | 1 | 4
Infective tenosynovitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 3
Intervertebral discitis (Infections and infestations) | 0 | 1
Intestinal gangrene (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 2
Lobar pneumonia (Infections and infestations) | 7 | 5
Localised infection (Infections and infestations) | 5 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 2 | 1
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Neuroborreliosis (Infections and infestations) | 1 | 1
Oral viral infection (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 6 | 6
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1
Periorbital cellulitis (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 105 | 73
Pneumonia bacterial (Infections and infestations) | 3 | 0
Pneumonia haemophilus (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 2 | 0
Post procedural infection (Infections and infestations) | 4 | 1
Postoperative abscess (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 2 | 5
Psoas abscess (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 6 | 10
Pyelonephritis acute (Infections and infestations) | 0 | 1
Pyothorax (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Salmonella sepsis (Infections and infestations) | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 2
Scrotal infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 14 | 20
Sepsis syndrome (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 1 | 1
Staphylococcal abscess (Infections and infestations) | 2 | 2
Staphylococcal bacteraemia (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 4 | 6
Staphylococcal osteomyelitis (Infections and infestations) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 2
Tooth infection (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 25 | 21
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 8 | 10
Viral infection (Infections and infestations) | 2 | 3
Viral labyrinthitis (Infections and infestations) | 0 | 1
Viral myocarditis (Infections and infestations) | 1 | 0
Vulval abscess (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 2 | 4
Wound infection pseudomonas (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 2
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1
Accidental exposure (Injury, poisoning and procedural complications) | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 2
Anaesthetic complication neurological (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 15 | 7
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 3 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 4
Device failure (Injury, poisoning and procedural complications) | 2 | 2
Device migration (Injury, poisoning and procedural complications) | 0 | 1
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 3
Excoriation (Injury, poisoning and procedural complications) | 1 | 1
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Failure of implant (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 13 | 13
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 | 4
Femur fracture (Injury, poisoning and procedural complications) | 9 | 5
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 1
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 1
Graft dysfunction (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 3 | 2
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 2
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 22 | 20
Humerus fracture (Injury, poisoning and procedural complications) | 7 | 6
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 1 | 0
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 2 | 3
Injury (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 4 | 0
Joint injury (Injury, poisoning and procedural complications) | 3 | 1
Kidney rupture (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 3 | 3
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 4
Lung injury (Injury, poisoning and procedural complications) | 0 | 1
Medical device complication (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 3
Multiple injuries (Injury, poisoning and procedural complications) | 2 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Neck injury (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Pacemaker complication (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 2 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 4 | 2
Pneumonitis chemical (Injury, poisoning and procedural complications) | 1 | 0
Pocket erosion (Injury, poisoning and procedural complications) | 1 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 0 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 2
Pubic rami fracture (Injury, poisoning and procedural complications) | 0 | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 9
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 2
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 3
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 1
Stent occlusion (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 6 | 13
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Surgical procedure repeated (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 5
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 3 | 4
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 2
Traumatic brain injury (Injury, poisoning and procedural complications) | 2 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 6 | 6
Urethral stricture postoperative (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 3
Wound complication (Injury, poisoning and procedural complications) | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 6 | 1
Band neutrophil count increased (Investigations) | 0 | 1
Biopsy liver (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 2
Blood glucose abnormal (Investigations) | 0 | 1
Blood glucose decreased (Investigations) | 1 | 0
Blood glucose fluctuation (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 3 | 4
Blood potassium decreased (Investigations) | 2 | 0
Blood potassium increased (Investigations) | 0 | 1
Blood pressure decreased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 2 | 1
Blood pressure orthostatic decreased (Investigations) | 1 | 0
Blood sodium decreased (Investigations) | 1 | 1
Cardiac murmur (Investigations) | 0 | 1
Cardiac stress test abnormal (Investigations) | 0 | 1
Cardiac stress test normal (Investigations) | 0 | 1
Cardioactive drug level increased (Investigations) | 1 | 0
Chest X-ray abnormal (Investigations) | 1 | 0
Coagulation test abnormal (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Heart rate decreased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 0 | 1
Heart rate irregular (Investigations) | 1 | 2
Hepatic enzyme increased (Investigations) | 2 | 1
International normalised ratio increased (Investigations) | 3 | 1
Liver function test abnormal (Investigations) | 1 | 0
Occult blood positive (Investigations) | 2 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Red blood cell count increased (Investigations) | 1 | 0
Scan myocardial perfusion abnormal (Investigations) | 1 | 1
Transaminases increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 1 | 1
Urine output decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 0
Weight increased (Investigations) | 0 | 2
White blood cell count increased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 39 | 51
Diabetes mellitus (Metabolism and nutrition disorders) | 13 | 18
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 7 | 5
Diabetic foot (Metabolism and nutrition disorders) | 5 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 4 | 5
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 3
Failure to thrive (Metabolism and nutrition disorders) | 1 | 2
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 3 | 7
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 10 | 11
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 32 | 24
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 17
Hypovolaemia (Metabolism and nutrition disorders) | 5 | 3
Ketosis (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0
Overweight (Metabolism and nutrition disorders) | 0 | 1
Podagra (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 12
Arthritis (Musculoskeletal and connective tissue disorders) | 12 | 10
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 18
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone erosion (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 7 | 4
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 3
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 9 | 11
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 13 | 7
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 41 | 58
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 4
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 7 | 5
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 11 | 11
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 | 2
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 2
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 6
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 9
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bone sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 | 14
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 18
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gliosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 22
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant lymphoid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 6
Malignant neoplasm of islets of Langerhans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Oropharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Penile malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 38 | 51
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Refractory anaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sebaceous adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Alcoholic seizure (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0
Anoxic encephalopathy (Nervous system disorders) | 2 | 0
Ataxia (Nervous system disorders) | 0 | 3
Balance disorder (Nervous system disorders) | 0 | 1
Brain mass (Nervous system disorders) | 0 | 2
Carotid artery disease (Nervous system disorders) | 5 | 4
Carotid artery occlusion (Nervous system disorders) | 2 | 4
Carotid artery stenosis (Nervous system disorders) | 27 | 26
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 2 | 1
Cerebral artery occlusion (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 3 | 8
Cerebral infarction (Nervous system disorders) | 6 | 7
Cerebral ischaemia (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 86 | 88
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1
Cervical cord compression (Nervous system disorders) | 0 | 1
Cervical myelopathy (Nervous system disorders) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 2 | 2
Convulsion (Nervous system disorders) | 2 | 7
Critical illness polyneuropathy (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 4 | 2
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Diabetic hyperosmolar coma (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 18 | 31
Dizziness postural (Nervous system disorders) | 1 | 2
Drop attacks (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 1
Dystonia (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 2
Epilepsy (Nervous system disorders) | 1 | 2
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Facial palsy (Nervous system disorders) | 1 | 3
Global amnesia (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 9
Hemiparesis (Nervous system disorders) | 4 | 5
Hemiplegia (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 1
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 4 | 5
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Hypokinesia (Nervous system disorders) | 1 | 0
Hypoxic encephalopathy (Nervous system disorders) | 1 | 1
Intracranial aneurysm (Nervous system disorders) | 3 | 0
Intracranial hypotension (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 2
Ischaemic stroke (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 2
Loss of consciousness (Nervous system disorders) | 2 | 3
Lumbar radiculopathy (Nervous system disorders) | 0 | 2
Metabolic encephalopathy (Nervous system disorders) | 2 | 0
Monoplegia (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 2 | 1
Myelopathy (Nervous system disorders) | 2 | 0
Narcolepsy (Nervous system disorders) | 1 | 0
Nerve root compression (Nervous system disorders) | 1 | 1
Nerve root lesion (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 2 | 0
Partial seizures (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 16 | 15
Radiculopathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 2 | 3
Simple partial seizures (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 3 | 3
Subdural hygroma (Nervous system disorders) | 0 | 1
Supranuclear palsy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 51 | 76
Syncope vasovagal (Nervous system disorders) | 3 | 1
Tarsal tunnel syndrome (Nervous system disorders) | 0 | 1
Thalamic infarction (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 52 | 52
Tremor (Nervous system disorders) | 1 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
VIth nerve paralysis (Nervous system disorders) | 2 | 0
Vascular dementia (Nervous system disorders) | 0 | 1
Vertebral artery stenosis (Nervous system disorders) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Perineal laceration (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 1
Agitated depression (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 2 | 0
Alcoholism (Psychiatric disorders) | 4 | 1
Anxiety (Psychiatric disorders) | 4 | 5
Anxiety disorder (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 6 | 5
Crying (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 2 | 5
Depression suicidal (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 1
Generalised anxiety disorder (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 1
Intentional self-injury (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 2
Mania (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 8 | 4
Panic attack (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 1
Restlessness (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 2
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 2
Azotaemia (Renal and urinary disorders) | 1 | 2
Bladder disorder (Renal and urinary disorders) | 1 | 1
Bladder neck obstruction (Renal and urinary disorders) | 0 | 2
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Bladder perforation (Renal and urinary disorders) | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 3
Bladder spasm (Renal and urinary disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 3 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 2
Calculus urethral (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 3 | 2
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 7 | 9
Hydronephrosis (Renal and urinary disorders) | 2 | 2
Hypertonic bladder (Renal and urinary disorders) | 1 | 0
Microalbuminuria (Renal and urinary disorders) | 3 | 1
Nephrolithiasis (Renal and urinary disorders) | 5 | 5
Nephrosclerosis (Renal and urinary disorders) | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Pyuria (Renal and urinary disorders) | 0 | 1
Renal aneurysm (Renal and urinary disorders) | 0 | 1
Renal artery arteriosclerosis (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 7 | 9
Renal disorder (Renal and urinary disorders) | 3 | 3
Renal failure (Renal and urinary disorders) | 30 | 45
Renal failure acute (Renal and urinary disorders) | 32 | 38
Renal failure chronic (Renal and urinary disorders) | 6 | 8
Renal impairment (Renal and urinary disorders) | 2 | 3
Renal mass (Renal and urinary disorders) | 4 | 3
Renal tubular necrosis (Renal and urinary disorders) | 2 | 1
Stag horn calculus (Renal and urinary disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 7 | 8
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 13 | 11
Breast mass (Reproductive system and breast disorders) | 0 | 1
Colpocele (Reproductive system and breast disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 2 | 2
Ovarian mass (Reproductive system and breast disorders) | 1 | 1
Pelvic prolapse (Reproductive system and breast disorders) | 1 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0
Prostatism (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 3 | 3
Prostatomegaly (Reproductive system and breast disorders) | 0 | 2
Rectocele (Reproductive system and breast disorders) | 2 | 1
Uterine prolapse (Reproductive system and breast disorders) | 2 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Allergic respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 42 | 49
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 | 43
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Laryngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 15 | 9
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 14 | 28
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 18 | 12
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 7 | 13
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 6
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Cardiac assistance device user (Social circumstances) | 0 | 1
Joint prosthesis user (Social circumstances) | 2 | 0
Penile prosthesis user (Social circumstances) | 1 | 0
Arterial bypass operation (Surgical and medical procedures) | 0 | 1
Coronary revascularisation (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1
Angiopathy (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 13 | 21
Aortic aneurysm rupture (Vascular disorders) | 1 | 2
Aortic dilatation (Vascular disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Aortic intramural haematoma (Vascular disorders) | 0 | 1
Aortic rupture (Vascular disorders) | 1 | 1
Aortic stenosis (Vascular disorders) | 5 | 8
Arterial insufficiency (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 7 | 8
Arterial restenosis (Vascular disorders) | 0 | 1
Arterial stenosis (Vascular disorders) | 1 | 4
Arterial thrombosis (Vascular disorders) | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 0 | 2
Arteriosclerosis (Vascular disorders) | 11 | 14
Arteriosclerosis obliterans (Vascular disorders) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 1 | 0
Blood pressure inadequately controlled (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 14 | 15
Embolism (Vascular disorders) | 1 | 1
Essential hypertension (Vascular disorders) | 1 | 0
Femoral arterial stenosis (Vascular disorders) | 2 | 3
Femoral artery aneurysm (Vascular disorders) | 1 | 1
Femoral artery occlusion (Vascular disorders) | 0 | 6
Haematoma (Vascular disorders) | 2 | 3
Haemorrhage (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 10 | 23
Hypertensive crisis (Vascular disorders) | 1 | 11
Hypertensive emergency (Vascular disorders) | 0 | 1
Hypoperfusion (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 22 | 30
Hypovolaemic shock (Vascular disorders) | 0 | 2
Iliac artery occlusion (Vascular disorders) | 2 | 1
Iliac artery stenosis (Vascular disorders) | 4 | 3
Infarction (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 4 | 16
Ischaemia (Vascular disorders) | 2 | 3
Labile hypertension (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 0 | 1
Orthostatic hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 5 | 15
Peripheral arterial occlusive disease (Vascular disorders) | 8 | 2
Peripheral artery aneurysm (Vascular disorders) | 3 | 4
Peripheral embolism (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 3 | 5
Peripheral vascular disorder (Vascular disorders) | 21 | 27
Phlebitis (Vascular disorders) | 0 | 1
Poor peripheral circulation (Vascular disorders) | 1 | 0
Post thrombotic syndrome (Vascular disorders) | 1 | 0
Renovascular hypertension (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 0 | 1
Subclavian steal syndrome (Vascular disorders) | 1 | 0
Takayasu's arteritis (Vascular disorders) | 0 | 1
Temporal arteritis (Vascular disorders) | 0 | 2
Thrombophlebitis (Vascular disorders) | 0 | 3
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 3 | 3
Varicose vein (Vascular disorders) | 1 | 0
Vascular occlusion (Vascular disorders) | 2 | 0
Vascular pseudoaneurysm (Vascular disorders) | 2 | 1
Vascular stenosis (Vascular disorders) | 1 | 1
Venous occlusion (Vascular disorders) | 1 | 0
Venous stasis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Benazepril / Amlodipine (N=5740) | Benazepril / HCTZ (N=5757)
Oedema peripheral (General disorders) | 1787 | 768
Dizziness (Nervous system disorders) | 1175 | 1440
Cough (Respiratory, thoracic and mediastinal disorders) | 1172 | 1217

LIMITATIONS AND CAVEATS:
Study was stopped early, as recommended by the Data Monitoring Committee, due to positive efficacy results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.